CLINICAL TRIAL: NCT02338245
Title: Randomized Phase 2A/2B Study to Compare the Efficacy and Safety of ASLAN001 + Capecitabine to Lapatinib + Capecitabine in Patients With HER 2-Positive MBC That Has Failed on Prior Trastuzumab Therapy
Brief Title: Study of ASLAN001 in Combination With Capecitabine in MBC That Has Failed on Prior Trastuzumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ASLAN Pharmaceuticals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASLAN001-003
Record Dates: First submitted 2015-01-06; First posted 2015-01-14 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Arm A (Experimental): ASLAN001 + Capecitabine
  Interventions: Drug: ASLAN001; Drug: Capecitabine
- Treatment Arm B (Active Comparator): Lapatinib + Capecitabine
  Interventions: Drug: Lapatinib; Drug: Capecitabine

INTERVENTIONS:
Drug: ASLAN001 — ASLAN001 400mg BID
  Arms: Treatment Arm A
Drug: Lapatinib — Lapatinib 1250mg QD
  Other Names: Tykerb
  Arms: Treatment Arm B
Drug: Capecitabine — Capecitabine 1000mg/kg BID days 1-14 of a 21-day cycle
  Other Names: Xeloda

SUMMARY:
This is an open-label, randomized, parallel group Phase 2A/2B study to evaluate the clinical activity of ASLAN001 in combination with capecitabine compared with lapatinib in combination with capecitabine in patients with HER2 positive metastatic breast cancer that has failed on prior trastuzumab therapy.

DETAILED DESCRIPTION:
Phase 2A Design:

The Phase 2A part is an open-label, randomized, parallel group study using tumor size as its primary efficacy endpoint. Approximately 44 eligible patients will be randomized in a 1:1 ratio to receive either ASLAN001 400 mg orally twice daily (BID) or lapatinib 1250 mg orally once daily (QD), both on a background of capecitabine 1000 mg/m2 orally BID for Days 1-14 of a 21-day cycle. Radiological imaging to assess disease status will be performed at baseline and every 6 weeks until disease progression (as assessed by the Investigator). Patients who have not experienced disease progression after 12 weeks may continue to receive randomized therapy and will continue to have radiological scans every 6 weeks until disease progression.

Criteria to Proceed to Phase 2B:

In the absence of any safety or tolerability concerns, continuation to the Phase 2B part of the study will be primarily based on the statistical comparison of the percentage change in tumor size from baseline to Week 12 and a one-sided p-value <0.1 in favor of the ASLAN001-containing treatment arm would be supportive of continuation to Phase 2B.

Phase 2B Design:

The Phase 2B part of the study will continue to recruit if the pre-specified efficacy criteria are met in the Phase 2A part and if the tolerability of ASLAN001 in combination with capecitabine is considered acceptable.

The Phase 2B part is an open-label, randomized, parallel group study. In this part, approximately 160 patients will be randomized in a 1:1 ratio to receive either ASLAN001 400 mg BID or lapatinib 1250 mg QD, both in combination with capecitabine 1000 mg/m2 BID for Days 1-14 of a 21-day cycle.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented histological confirmation of breast cancer with HER 2 overexpression or gene amplification prior to study entry.
* Patients with HER 2-positive metastatic breast cancer that have failed on prior first line treatment with trastuzumab or who have progressed within 1 year of treatment with trastuzumab in adjuvant setting.
* Presence of at least one radiographically measurable disease (bone metastases and ascites are not considered measurable lesions).
* Patients of the respective country's legal age or older at the time of written informed consent.
* Patients with acceptable organ and hematological function

Exclusion Criteria:

* Patients with radiation treatment or major surgical procedures within 21 days prior to study entry.
* Patients with malabsorption syndrome, diseases significantly affecting gastrointestinal function, resection of the stomach or small bowel, or difficulty in swallowing and retaining oral medications.
* Patients with an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, unstable angina pectoris, cardiac arrhythmia, diabetes, hypertension, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with any history of other malignancy unless in remission for more than 1 year. (Nonmelanoma skin carcinoma and carcinoma-in-situ of uterine cervix treated with curative intent is not exclusionary).
* Patients with symptomatic central nervous system metastasis and/or on systemic steroids or anticonvulsants within 3 months before the first dose of randomized therapy.
* Patients who are pregnant or breast-feeding.
* Patients who were previously treated with ASLAN001 and/or with lapatinib.
* Patients who have received more than 2 lines of any therapies in metastatic stage.
* Patients who have received any investigational drug (or have used an investigational device) within 21 days or received any antineoplastic monoclonal antibodies within a period of 5 half-lives before receiving the first dose of randomized therapy.
* Patients with unresolved or unstable serious toxicity from prior administration of another investigational drug and/or prior cancer treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-12-29 (Actual); Primary Completion 2016-05-19 (Actual); Study Completion 2016-08-25 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy of ASLAN001 in combination with capecitabine, to lapatinib in combination with capecitabine in the percentage change from baseline tumor size at Week 12 | Week 12

SECONDARY OUTCOMES:
Safety for all metastatic breast cancer (MBC) subjects (Physical examination, body weight, vital signs, ECG parameter, hematology, clinical laboratory tests and Adverse Events) | estimated 2 years
  Physical exam, body weight, vital signs (Blood pressure, respiratory rate and body temperateure), ECG parameter, hematology, clinical laboratory tests (clinical chemistry, coagulation and urinalysis) and Adverse Events (AEs)/ Serious Adverse Events (SAEs)
To further compare the efficacy of ASLAN001 in combination with capecitabine to lapatinib in combination with capecitabine, as measured by PFS and tumor volume | Week 12
To further compare the efficacy of ASLAN001 in combination with capecitabine to lapatinib in combination with capecitabine, as measured by the Objective Response Rate (ORR), Duration of Response (DoR), and Overall Survival (OS) | 2 years
  Composite outcome measures

CONTACTS AND LOCATIONS:
Locations (12):
- Australia, Western Australia, Australia
- Hong Kong, Hong Kong, Hong Kong
- New Zealand (2):
  - New Zealand, Christchurch
  - New Zealand, Tauranga
- Philippines (2):
  - Philippines, Bacolod City
  - Philippines, Dasmariñas
- Singapore, Singapore, Singapore
- South Korea, Seoul, South Korea
- Taiwan (4):
  - Taiwan, Linkou District, Taoyuan
  - Taiwan, Kaohsiung City
  - Taiwan, Taichung
  - Taiwan, Taipei